CLINICAL TRIAL: NCT00554385
Title: The Long-term Safety and Tolerability of ABT-089 in Children With Attention-Deficit/Hyperactivity Disorder (ADHD): An Open-Label Extension Study
Brief Title: A Safety and Tolerability Study of ABT-089 in Children With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-178
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — pozanicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ABT-089

INTERVENTIONS:
Drug: ABT-089 — Up to 4 capsules will be taken once daily for 12 months. Dosage forms include 1 mg, 5 mg, 10 mg capsules and 40 mg tablets. Highest dose allowed is 80 mg per day.

SUMMARY:
The objective of this study is to evaluate the long-term safety and tolerability of ABT-089 in children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* The subject was randomized into Base Study (M06-888 or M10-345) and completed the Treatment Period.
* If female, subject must be practicing at least one method of birth control throughout the study.
* If female, the result of a pregnancy test is negative.
* The subject is judged to be in generally good health.

Exclusion Criteria:

* The subject experienced a serious adverse event in Base Study (M06-888 or M10-345) that the investigator considered "possibly" or "probably related" to study drug.
* The subject has taken any ADHD medication between the last dose of study drug in Study M06-888 or M10-345 and the first dose of study drug in the current study.
* The subject has a positive urine drug screen for alcohol or drugs of abuse.
* The subject anticipates a move outside the geographic area.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 283 (Actual)
Dates: Start 2007-11; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
ADHD-RS-IV (HV) | Day -1, Day 14, Months 1, 2, 3, 6, 9 & 12
CGI-ADHD-S | Day -1, Day 14, Months 1, 2, 3, 6, 9 & 12

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gault, M.D., Ph.D., Study Director — Abbott
Locations (23):
- United States (23):
  - Site Ref #/Investigator 6800, Little Rock, Arkansas
  - Site Ref #/Investigator 6812, Boulder, Colorado
  - Site Ref #/Investigator 8366, Bradenton, Florida
  - Site Ref #/Investigator 6808, Jacksonville, Florida
  - Site Ref #/Investigator 6827, Orlando, Florida
  - Site Ref #/Investigator 8383, Libertyville, Illinois
  - Site Ref #/Investigator 6802, Northbrook, Illinois
  - Site Ref #/Investigator 6824, Overland Park, Kansas
  - Site Ref #/Investigator 8428, Troy, Michigan
  - Site Ref #/Investigator 6902, Omaha, Nebraska
  - Site Ref #/Investigator 6856, Las Vegas, Nevada
  - Site Ref #/Investigator 6683, Clementon, New Jersey
  - Site Ref #/Investigator 8297, Oklahoma City, Oklahoma
  - Site Ref #/Investigator 6682, Eugene, Oregon
  - Site Ref #/Investigator 6811, Portland, Oregon
  - Site Ref #/Investigator 8701, Portland, Oregon
  - Site Ref #/Investigator 6681, Salem, Oregon
  - Site Ref #/Investigator 6799, Charleston, South Carolina
  - Site Ref #/Investigator 7955, Memphis, Tennessee
  - Site Ref #/Investigator 6836, Austin, Texas
  - Site Ref #/Investigator 6835, Herndon, Virginia
  - Site Ref #/Investigator 6791, Bellevue, Washington
  - Site Ref #/Investigator 6838, Middleton, Wisconsin